CLINICAL TRIAL: NCT00302536
Title: Tacrolimus Treatment of Patients With Idiopathic Focal Segmental
Brief Title: Tacrolimus Treatment of Patients With Idiopathic Focal Segmental Glomerulosclerosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was less patients recruited.
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0604
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2010-09

CONDITIONS: Focal Glomerulosclerosis
Keywords: Idiopathic Focal Segmental Glomerulosclerosis; Treatment; Steroids
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus
  Other Names: Tacrolimus, Prograf

SUMMARY:
The purpose of this study is to assess the efficacy of Tacrolimus Treatment of patients with idiopathic focal segmental glomerulosclerosis.

DETAILED DESCRIPTION:
Primary FSGS is a leading cause of end stage renal disease in adults, with complete loss of kidney function in 50% of patients over 10 years. Steroids, which are currently used to treat the disease, are effective in part of patients. Over the past decade, a number of studies have reported therapeutic efficacy for treatment with Cyclosporine-A (CSA) in patients with FSGS. Recent studies suggest that immunosuppressive therapy targeted against the calcineurin pathway of T-helper cells, for example, tacrolimus, may be effective in the treatment of primary FSGS. The experience with Tacrolimus (FK506) in the treatment of patients with FSGS has been limited to uncontrolled trials in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-50 years at onset of signs or symptoms of FSGS
* Biopsy proven FSGS
* Estimated glomerular filtration rate (GFR) ≥ 40 ml/min/1.73 m2
* Urine protein > 3.5 g/24h
* Biopsy confirmed primary FSGS (including all subtypes)
* Willingness to follow the clinical trial protocol, including medications, and baseline and follow-up visits and procedures

Exclusion Criteria:

* Secondary FSGS
* Prior therapy with sirolimus, CSA, MMF, or azathioprin, cytoxan, chlorambucil levamisole, methotrexate, or nitrogen mustard in the last 90 days
* Active/serious infection
* Malignancy
* Previously diagnosed diabetes mellitus type 1 or 2
* Clinical evidence of cirrhosis or chronic active liver disease
* History of significant gastrointestinal disorder
* Allergy to study medications, and Inability to consent/assent

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2010-05 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of Tacrolimus Treatment Idiopathic Focal Segmental Glomerulosclerosis | 18 months

SECONDARY OUTCOMES:
To investigate the safety and tolerability of Tacrolimus vs Steroids in Treatment Idiopathic Focal Segmental Glomerulosclerosis | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-hong Liu, M.D., Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732